CLINICAL TRIAL: NCT00635973
Title: Multi-Centre, Open-Label Extension Trial of Treatment With ZD1839 (Iressa) in Patients Who Have Been Treated in Other ZD1839 Clinical Trials and May Benefit From Continued Monotherapy ZD 1839.
Brief Title: Open-Label Extension of Other SZ1839 (Iressa) Trials
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Alison Armour Medical Science Director, AstraZeneca
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1839IL/0026; D7913C00026
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Last update posted 2009-04-22 (Estimated); Status verified 2009-04

CONDITIONS: Cancer
Keywords: Iressa; Gefitinib; Cancer; Patients diagnosed with cancer who have previously received Iressa in an Iressa clinical trial
MeSH Terms: conditions — Neoplasms | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Gefitinib (Iressa) — Iressa

SUMMARY:
A trial to assess patients who have been treated with Iressa in a previous clinical trial and may benefit from continued treatment with Iressa.

ELIGIBILITY:
Inclusion Criteria:

* Received treatment in a previous Iressa clinical trial
* Provided Informed Consent to participate in the trial
* 30 days or less since completing the previous Iressa trial.

Exclusion Criteria:

* Radiotherapy completed more than 14 days before starting treatment in this trial
* Incomplete healing from prior surgery
* Withdrawal from previous Iressa trial due to unacceptable toxicity to major organs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2000-02; Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Every 28 days

SECONDARY OUTCOMES:
Progression Free Survival | Every 28 days
Survival | Every 28 days